CLINICAL TRIAL: NCT04609800
Title: CAROLINE: An Observational, Prospective, Multicenter Study, on the Utilization of Cabozantinib in Adult Patients With Advanced or Metastatic Renal Cell Carcinoma (RCC) in 2nd Line Treatment Following Prior Vascular Endothelial Growth Factor (VEGF)-Targeted Therapy Under Real-real Life Clinical Setting in France.
Brief Title: Study on the Utilization of Cabozantinib in Adult Patients With Advanced or Metastatic Renal Cell Carcinoma (RCC) in 2nd Line Treatment Following Prior Vascular Endothelial Growth Factor (VEGF)-Targeted Therapy Under Real-real Life Clinical Setting in France.
Acronym: CAROLINE
Status: Withdrawn | Type: Observational
Why Stopped: Unfavorable opinion of IRB/IEC
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-FR-60000-070
Record Dates: First submitted 2020-10-07; First posted 2020-10-30 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma (clear cell or non-clear cell)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the protocol is to assess the Overall Survival (OS) at 1 year in patients after cabozantinib initiation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 age at the time of cabozantinib initiation
* Pathologically confirmed diagnosis of Renal Cell Carcinoma (Clear Cell or non-Clear Cell) cancer considered as advanced or metastatic at the time of cabozantinib initiation
* Intention to be treated with cabozantinib tablets according to the current local Summary of Product Characteristics (SmPC) (France)
* Initiating cabozantinib as a second line of treatment (Baseline visit must be performed before cabozantinib first intake)

Exclusion Criteria:

* He/she is already included in an interventional trial with an investigational product at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data of 195 participants suffering from advanced or metastatic RCC and treated with cabozantinib will be collected. During the study, two questionnaires (FKSI 19 and BPI-SF) will be filled in by patients.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11-06 (Estimated); Primary Completion 2023-05-10 (Estimated); Study Completion 2023-05-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) rate at 1 year after cabozantinib initiation | up to 12 months
  OS is the time between treatment initiation and the date of death from any cause. For participants who are alive, their survival time will be censored at the last date that they were known to be alive if before 1 year.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) at 1 year | Day 15, 1 month, 3, 6 and 12 months
  ORR is defined as the proportion of participants who achieve partial or complete response from the start of the study treatment. The ORR will be assessed by tumour response evaluation according to investigator assessment. Tumour response will be evaluated per routine clinical practice by the physician.
Best Overall Response (BOR) at 1 year | Day 15, 1 month, 3, 6 and 12 months
  BOR is the best response recorded from the start of the study treatment until the disease progression/recurrence. The BOR will be assessed by tumour response evaluation according to investigator assessment. Tumour response will be evaluated per routine clinical practice by the physician.
Progression Free Survival (PFS) at 1 year | Day 15, 1 month, 3, 6 and 12 months
  PFS is defined as the time elapsed from the date of first treatment intake to the date of documented progression reported by the investigator or death due to any cause, whichever occurs first. Disease progression will be assessed by tumour response evaluation according to investigator assessment. Tumour response will be evaluated per routine clinical practice as Progressive / not progressive disease by the physician.
Previous systemic neoadjuvant and adjuvant therapies for RCC prior cabozantinib initiation in terms of nature of the therapy, duration, and reason for discontinuation. | Baseline
First-line therapy for RCC prior cabozantinib initiation in terms of nature of the therapy, duration, and reason for discontinuation. | Baseline
Pattern of use of cabozantinib | Baseline, day 15, 1 month, 3, 6 and 12 months
  Dose modification, reason of modification and treatment duration of cabozantinib will be described from cabozantinib initiation until participants' end of study treatment or study withdrawal.
Quality of life (QoL) change according to Functional Assessment of Cancer Therapy (FKSI-19) questionnaire | Baseline, day 15, 1 month, 3, 6 and 12 months
  QoL change from baseline. The score will be evaluated with FKSI 19 questionnaires at the planned visits and at treatment discontinuation. The FKSI-19 is a disease-specific instrument that measures disease and treatment-related symptoms in 4 domains by using a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). Higher scores represent better health. A negative change from Baseline represents a worsening of condition.
Pain assessment | Baseline, day 15, 1 month, 3, 6 and 12 months
  To assess pain according to the Brief Pain Inventory-Short Form (BPI-SF) questionnaire and analgesic consumption/duration and the time for improvement of symptomatology. BPI-SF has a scale of 0 to 10 with 0 indicating "No pain" and 10 indicating "Pain as bad as you can imagine".
Subsequent systemic treatment for RCC after cabozantinib discontinuation in terms of the description of the nature of the therapy, starting date. | End of Study visit (12 months if the patient didn't discontinue earlier)
Safety of cabozantinib in the real-world setting | Day 15, 1 month, 3, 6 and 12 months
  Incidence of Adverse Events (AEs),Serious Adverse Events (SAEs) assessed overall and by intensity and causality.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen